CLINICAL TRIAL: NCT01172782
Title: The Analgesic Effect of Intrathecal Hydromorphone Injection on Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Korea University (Other)
Responsible Party: Too Jae Min, anesthesiology department, clinical professor, Department of Anesthesiology and Pain Medicine, Korea University Ansan Hospital, Korea University College of Medicine, Ansan, Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: minware2
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-01

CONDITIONS: Pain Measurement; Visual Analog Pain Scale
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control group (Placebo Comparator): control group (CG) received 6 mg of hyperbaric bupivacaine and 0.05 mL of saline.
  Interventions: Drug: Hydromorphone
- 2.5 ug hydromorphone recieved group (Active Comparator): the 2.5 μg hydromorphone group (2.5HG) received 1.2 (6 mg) mL of 0.5% hyperbaric bupivacaine and 2.5 μg of hydromorphone in 0.05 mL of saline
  Interventions: Drug: Hydromorphone
- 5 μg hydromorphone group (Active Comparator): 5 μg hydromorphone group received 1.2 mL of 0.5% hyperbaric bupivacaine and 5 μg of hydromorphone in 0.05 mL of saline
  Interventions: Drug: Hydromorphone
- the 10 μg hydromorpnone group (Active Comparator): the 10 μg hydromorphone group received 1.2 mL of 0.5% hyperbaric bupivacaine and 10 μg of hydromorphone in 0.05 mL of saline.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — 2.5, 5, 10 ug of hydromorphone, intrathecal injection, single injection. duration of intrathecal injection are not fully studied.

SUMMARY:
The purpose of this study is to evaluate the adequate dose of intrathecal hydromorphone injection for postoperative pain relief after knee arthroscopic surgery.

DETAILED DESCRIPTION:
Sixty patients who were undergoing unilateral knee arthroscopy randomly received unilateral spinal anesthesia with 0.5% hyperbaric bupivacaine 6 mg combined with normal saline 0.05 mL or hydromorphone 2.5, 5 or, 10 μg/0.05 mL. The verbal numerical rating scale (VNRS) pain scores were measured at 30 minutes and 2, 4, 6, 12 and 24 hours postoperatively, and the side effects of hydromorphone were recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-II (age range: 18-72 years)
* Informed consent obtained patients

Exclusion Criteria:

* The exclusion criteria included evidence of neurological or neuromuscular disease, respiratory or cardiac disease, diabetes mellitus or peripheral neuropathy, as well as those patients who were receiving chronic analgesic therapy or who had infection at the intended site of spinal needle insertion or who had hypersensitivity to amide local anesthetics or opioids

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Visual Analgesic Numberic Score | during postoperative recovery period.

REFERENCES:
- [Derived] Lee YS, Park YC, Kim JH, Kim WY, Yoon SZ, Moon MG, Min TJ. Intrathecal hydromorphone added to hyperbaric bupivacaine for postoperative pain relief after knee arthroscopic surgery: a prospective, randomised, controlled trial. Eur J Anaesthesiol. 2012 Jan;29(1):17-21. doi: 10.1097/EJA.0b013e3283476055. PMID 21562420